CLINICAL TRIAL: NCT03244358
Title: Evaluation of Epalrestat in Metastatic Triple-negative Breast Cancer:A Single Arm,Single Center,Phase II Study
Brief Title: Evaluation of Epalrestat in Metastatic Triple-negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty accruing subjects the study accrual was closed
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, professer, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-010
Record Dates: First submitted 2017-07-23; First posted 2017-08-09 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Epalrestat
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — epalrestat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Epalrestat (Experimental): Epalrestat added to standard treatment
  Interventions: Drug: Epalrestat

INTERVENTIONS:
Drug: Epalrestat — Epalrestat 50mg tid added to standard chemotherapy treatment
  Other Names: Tanglin (Yangtze River Pharmaceutical Group), China

SUMMARY:
To evaluate the efficacy and safety of Epalrestat in the treatment of metastatic triple negative breast

DETAILED DESCRIPTION:
This is a phase II,single center,prospective, single arm clinical trials. The objective is to evaluate the efficacy and safetyof Epalrestat in the treatment of metastatic triple negative breast.Primary endpoint is 16-week clinical benefit rate (CBR).

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years, ≤70 years.
* Minimum life expectancy 16 weeks
* Histologicalconfirmation of hormone receptor negative and HER2 negative breast cancer(IHC:ER -, PR-) on primary tumour at diagnosis/on biopsy of metastasis
* Clinical or histological confirmation of metastatic or locally advanced disease not amenable to curative surgical resection
* ECOG 0-2 with no deterioration over previous 2 weeks Measurable disease
* Adequate bone marrow and organ function
* Availability of archival tumour sample or fresh biopsy Informed consent
* Normal organ function

Exclusion Criteria:

* Last dose chemotherapy, immunotherapy targeted therapy, biological therapy or tumour embolisation <21 days prior to study treatment
* Last dose of palliative radiotherapy <7 days prior to study treatment
* Rapidly progressive visceral disease not suitable for further therapy
* Spinal cord compression or brain/meningeal metastases unless asymptomatic, treated and stable and not requiring steroids for ≥ 4 weeks study treatment
* Major surgery (excluding placement of vascular access) within 4 weeks before study treatment
* Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and HIV
* With the exception of alopecia, any unresolved toxicities from previous therapy greater than CTCAE grade 1 before study treatment
* Elevated ALP in absence of bone metastasis
* Evidence of dementia, altered mental status or any psychiatric condition that would prohibit understanding or rendering of informed consent
* Participation in another study with investigational product during last 30 days
* Inability or unwillingness to comply with study procedures, including inability to take regular oral medication

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 30 months
  the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Overall Survival | 3 years
  OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: zhongyu yuan, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No